CLINICAL TRIAL: NCT03783000
Title: Investigation of Pharmacokinetics and Absolute Oral Bioavailability of BI 425809 Administered as an Oral Dose With an Intravenous Microtracer Dose of [C-14]-BI 425809 in Healthy Male Volunteers
Brief Title: A Study in Healthy Men to Measure the Amount of BI 425809 in the Blood When Taken as a Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1346-0015; 2018-001194-24 (EudraCT Number)
Record Dates: First submitted 2018-12-19; First posted 2018-12-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Healthy
MeSH Terms: interventions — BI 425809

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All subjects (Experimental): Treatment T followed by Treatment R
  Interventions: Drug: BI 425809; Drug: BI 425809 mixed with [C-14]-BI 425809

INTERVENTIONS:
Drug: BI 425809 — Treatment T
  Other Names: Iclepertin
Drug: BI 425809 mixed with [C-14]-BI 425809 — Treatment R
  Other Names: Iclepertin

SUMMARY:
The primary objective of this trial is to investigate the absolute oral bioavailability of BI 425809 administered as tablet (Test, T) compared to [C-14]-BI 425809 administered as intravenous microtracer (Reference, R).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, based on a complete medical history including a physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 65 years (incl.)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and local legislation
* Subjects who are sexually active must use, with their partner, highly effective contraception from the time of administration of trial medication until 4 months after administration of trial medication. Adequate methods are:

  * Condoms plus use of hormonal contraception by the female partner that started at least 2 months prior to administration of trial medication (e.g., implants, injectables, combined oral or vaginal contraceptives, intrauterine device) or
  * Condoms plus surgical sterilization (vasectomy at least 1 year prior to enrolment) or
  * Condoms plus surgically sterilised partner (including hysterectomy) or
  * Condoms plus intrauterine device or
  * Condoms plus partner of non-childbearing potential (including homosexual men) Subjects are required to use condoms to prevent unintended exposure of the partner to the study drug via seminal fluid.
  * Alternatively, true abstinence is acceptable when it is in line with the subject's preferred and usual lifestyle. If a subject is usually not sexually active but becomes active, with their partner, they must comply with the contraceptive requirements detailed above.

Exclusion Criteria:

* Any finding in the medical examination (including Blood Pressure (BP), Pulse Rate (PR) or Electrocardiogram (ECG)) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 139 mmHg, diastolic blood pressure outside the range of 45 to 89 mmHg, or pulse rate outside the range of 40 to 100 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Clinically significant gastrointestinal, hepatic, renal, respiratory (including but not limited to interstitial lung disease), cardiovascular, metabolic, immunological or hormonal disorders
* Further exclusion criteria apply

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2019-03-06 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ (area under the concentration-time curve of the analyte over the time interval from 0 to infinity) | Up to 168 hours

SECONDARY OUTCOMES:
Cmax (maximum measured concentration of the analyte in plasma) | Up to 168 hours

CONTACTS AND LOCATIONS:
Locations (1):
- PRA Health Sciences Onderzoekscentrum Martini, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). For more details refer to: http://trials.boehringer-ingelheim.com/

REFERENCES:
- [Derived] Burkard U, Desch M, Shatillo Y, Wunderlich G, Mack SR, Schlecker C, Teitelbaum AM, Liu P, Chan TS. The Absolute Bioavailability, Absorption, Distribution, Metabolism, and Excretion of BI 425809 Administered as an Oral Dose or an Oral Dose with an Intravenous Microtracer Dose of [14C]-BI 425809 in Healthy Males. Clin Drug Investig. 2022 Jan;42(1):87-99. doi: 10.1007/s40261-021-01111-9. Epub 2021 Dec 22. PMID 34936055